CLINICAL TRIAL: NCT01617109
Title: Optimizing Vitamin D Status During Initial Military Training: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Optimizing Vitamin D Status During Initial Military Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H12-09; 13-24HC
Record Dates: First submitted 2012-06-01; First posted 2012-06-12 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Bone Health; Nutrition Status
Keywords: Vitamin D; Calcium; Parathyroid hormone; Bone; Bone formation; Bone resorption; Micronutrients; Trace Elements
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo
- Ca/Vit D (Experimental)
  Interventions: Dietary Supplement: Ca/Vit D

INTERVENTIONS:
Dietary Supplement: Ca/Vit D — 800IU vitamin D3 and 2000mg elemental calcium (as calcium carbonate); administered as 5 pills daily or 2 snack bars
  Arms: Ca/Vit D
Other: Placebo — administered as 5 pills daily or as 2 snack bars
  Arms: Placebo

SUMMARY:
The primary objective of this randomized, double-blind, placebo-controlled trial is to determine the effect of vitamin D and calcium supplementation (800IU and 2000mg, respectively) on biochemical indicators of nutritional status and bone health in military personnel during Army basic combat training (BCT) and Air Force basic military training (BMT).

The investigators hypothesize that daily supplementation with vitamin D and calcium during military training will improve vitamin D status, stabilize PTH levels, and result in improvements in markers of bone health. As a result of the investigators study design, the findings will provide critically important data regarding the concentration of vitamin D in blood necessary to stabilize PTH levels and to optimize bone formation during initial military training.

DETAILED DESCRIPTION:
Vitamin D is an essential nutrient for maintaining bone health. Previous work from our laboratory indicates that vitamin D status may decline in Soldiers during BCT, even during the summer months in the Southeastern United States. Stress fractures may affect up to 5% of male and 21% of female Soldiers during training, resulting in attrition in up to 60% of affected personnel, but a recent report indicates that vitamin D and calcium supplementation may attenuate stress fracture risk by up to 20% in female Navy recruits. However, biochemical measures of nutritional status and associated markers of bone health were not collected in that study, leaving questions regarding the vitamin D and calcium requirements for military personnel during periods of elevated bone turnover.

ELIGIBILITY:
Inclusion Criteria:

* Female or male US Army or US Air Force Recruits
* Participating in Basic Combat Training or Basic Military Training, respectively

Exclusion Criteria:

* Pregnant or breastfeeding
* History of kidney stones or kidney disease

Ages: 17 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 342 (Actual)
Dates: Start 2012-06; Primary Completion 2014-01 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
Serum PTH pg/ml | Participants will be followed for the duration of basic combat training or basic military training, which are 7-9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James P McClung, Ph.D., Principal Investigator — US Army Research Institute of Environmental Medicine
Locations (2):
- United States (2):
  - Fort Sill, Fort Sill, Oklahoma
  - Lackland Air Force Base, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Andersen NE, Karl JP, Cable SJ, Williams KW, Rood JC, Young AJ, Lieberman HR, McClung JP. Vitamin D status in female military personnel during combat training. J Int Soc Sports Nutr. 2010 Dec 14;7:38. doi: 10.1186/1550-2783-7-38. PMID 21156069
- [Derived] Nakayama AT, Lutz LJ, Hruby A, Karl JP, McClung JP, Gaffney-Stomberg E. A dietary pattern rich in calcium, potassium, and protein is associated with tibia bone mineral content and strength in young adults entering initial military training. Am J Clin Nutr. 2019 Jan 1;109(1):186-196. doi: 10.1093/ajcn/nqy199. PMID 30615068
- [Derived] Lutz LJ, Gaffney-Stomberg E, Karl JP, Hughes JM, Guerriere KI, McClung JP. Dietary Intake in Relation to Military Dietary Reference Values During Army Basic Combat Training; a Multi-center, Cross-sectional Study. Mil Med. 2019 Mar 1;184(3-4):e223-e230. doi: 10.1093/milmed/usy153. PMID 29982620
- [Derived] Gaffney-Stomberg E, Lutz LJ, Rood JC, Cable SJ, Pasiakos SM, Young AJ, McClung JP. Calcium and vitamin D supplementation maintains parathyroid hormone and improves bone density during initial military training: a randomized, double-blind, placebo controlled trial. Bone. 2014 Nov;68:46-56. doi: 10.1016/j.bone.2014.08.002. Epub 2014 Aug 10. PMID 25118085